CLINICAL TRIAL: NCT02473432
Title: Neuromuscular Electroestimulation and Respiratory Muscle Training in the Management of Dysphagia of Subacute Stroke Patients
Brief Title: Neuromuscular Electroestimulation and Respiratory Muscle Training in Subacute Stroke
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Parc de Salut Mar (Other)
Responsible Party: Principal Investigator, Esther Marco Navarro, MD, Parc de Salut Mar
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PSM/RHB/NR/15
Record Dates: First submitted 2015-06-12; First posted 2015-06-16 (Estimated); Last update posted 2016-02-17 (Estimated); Status verified 2016-02

CONDITIONS: Dysphagia
Keywords: respiratory muscle training; neuromuscular electrical stimulation; oropharyngeal dysphagia; stroke; rehabilitation
MeSH Terms: conditions — Deglutition Disorders; Stroke | interventions — Breathing Exercises

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- RMT + usual care (Experimental): Device: Orygen-Dual® valve trainer Intensity: 30% of maximal respiratory pressures (increasing intervals: 10 cmH2O per week) Training schedule: 5 sets of 10 repetitions followed by 1-2 minutes of unloaded recovery breathing off the device, two sessions per day, 5 days per week, for 3 weeks.
  Interventions: Procedure: RMT + usual care
- NMES + usual care (Experimental): Device: Vital Stim (Chattanooga Group, Hixson, TN, USA) Administration of 80 Hz transcutaneous electrical biphasic stimulus Schedule: 40 minutes per day, 5 sessions per week during hospitalization in the Neurorehabilitation ward (3 weeks approx).
  Interventions: Procedure: NMES
- Usual care (Active Comparator): Usual care (standard multidisciplinary inpatient rehabilitation program) consisting of physical, occupational and speech therapy sessions to improve activities of daily life, mobility and communication skills (minimum 3 hours per day, 5 days a week, during 3 weeks), Standard swallow therapy (usual care of dysphagia in stroke patients) consists of physiotherapy, occupational therapy and speech therapy targeting specific swallow impairments. In the case of dysphagia, the standard pattern includes measures to protect the airway and compensatory techniques.
  Interventions: Procedure: Usual care

INTERVENTIONS:
Procedure: RMT + usual care — Respiratory muscle training is performed with the Orygen Dual valve (inspiratory and espiratory trainer)
  Other Names: Respiratory muscle training + usual care
  Arms: RMT + usual care
Procedure: NMES — Neuromuscular electrical stimulation is performed with the Vital Stim ® device (approved by the FDA for dysphagia treatment). It consists in the placement of two electrodes located in suprahyoid muscles as above described.
  Other Names: Neuromuscular electrical stimulation + usual care
  Arms: NMES + usual care
Procedure: Usual care — Standard swallow therapy consists of physiotherapy, occupational therapy and speech therapy targeting specific swallow impairments. In the case of dysphagia, the standard pattern includes measures to protect the airway and compensatory techniques.
  Other Names: Standard swallow therapy
  Arms: Usual care

SUMMARY:
This study, part of a larger research project (The Retornus Study), is aimed to evaluate new strategies to optimize rehabilitation outcomes in dysphagic stroke patients. Main objective is to assess effectiveness of neuromuscular electroestimulation (NMES) in combination with respiratory muscle training (RMT) in the treatment of oropharyngeal dysphagia in subacute stroke patients.

DETAILED DESCRIPTION:
Dysphagia is present in a significant proportion of subacute stroke patients (up to 85%, depending on the series) and is associated with an increase in medical complications such as bronchoaspirative pneumoniae which is responsible for approximately half of the deaths that occur in these patients. Besides, the risk of pneumonia in patients with dysphagia is three times higher compared to those patients without. Since there is no drug able to restore the swallowing and respiratory muscle function, neurological rehabilitation apperars to be as the mainstay of treatment of these disorders.

Respiratory muscle weakness is common after stroke, but how it contributes in the development of bronchoaspiration pneumonia is not well determined. In acute phases of stroke, the mechanism seems to be more related to an impaired central drive than the reduction of strength in respiratory muscle.

Otherwise, the NMES aims to improve muscle strength. The NMES accelerates swallowing recovery since it induces brain reorganitzation after stroke through sensory and motor stimulation of peripheral nerves, mainly in swallowing aerea.

ELIGIBILITY:
Inclusion Criteria:

* First-ever ischemic stroke
* Time since stroke onset: 1 to 3 weeks
* Tracheobronchial aspiration evaluated with the gold standard, videofluoroscopy,
* Cognitive impairment (Short Portable Mental Status Questionnaire less than 3)

Exclusion Criteria:

* Previous history of neurological diseases that might be associated with the presence of dysphagia
* Previous history of pulmonary diseases
* Significant alcohol abuse (>80 g/day) and 4) medical treatment with potential effect on muscle structure and function (steroids,thyroid hormones, immunosuppressors).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2013-12; Primary Completion 2015-06 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Penetration Aspiration Scale | up to 3 months follow-up
  Videofluoroscopy swallow assessment with the 8-point Penetration Aspiration Scale (PAS): PAS score of 1 indicates a normal test, scores from 2 to 5 indicate passage of material into the larynx that does not pass below the vocal folds (penetration) and scores from 6 to 8 indicate passage of material below the level of vocal folds (aspiration)

SECONDARY OUTCOMES:
Maximal inspiratory and expiratory muscle strength | up to 3 months follow-up
  Maximal respiratory muscle strength is assessed through maximal inspiratory and expiratory pressures (PImax and PEmax, respectively) measured at the mouth. To determine respiratory pressures, patients were urged to perform a maximum inspiration from residual volume against an occluded airway and a maximum expiratory effort from total lung capacity.
Security of swallowing oral phase | up to 3 months follow-up
  Security signs (tone of voice, coughing during or after eating, or desaturation of more than 3% compared to baseline pulse oximetry) are assessed with the Volume Viscosity Swallow Test:(V-VST).
Number of participants with signs of impaired efficacy ( Piecemeal deglutition and oropharyngeal residue). | up to 3 months follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Anna Guillen, MD, Principal Investigator — Parc de Salut Mar
Locations (1):
- Hospital de l'Esperança, Barcelona, Barcelona, Spain

REFERENCES:
- [Background] Wheeler KM, Chiara T, Sapienza CM. Surface electromyographic activity of the submental muscles during swallow and expiratory pressure threshold training tasks. Dysphagia. 2007 Apr;22(2):108-16. doi: 10.1007/s00455-006-9061-4. Epub 2007 Feb 10. PMID 17294298
- [Background] Huckabee ML, Doeltgen S. Emerging modalities in dysphagia rehabilitation: neuromuscular electrical stimulation. N Z Med J. 2007 Oct 12;120(1263):U2744. PMID 17972964
- [Background] Logemann JA. The effects of VitalStim on clinical and research thinking in dysphagia. Dysphagia. 2007 Jan;22(1):11-2. doi: 10.1007/s00455-006-9039-2. Epub 2007 Jan 10. No abstract available. PMID 17216392
- [Background] Martino R, Foley N, Bhogal S, Diamant N, Speechley M, Teasell R. Dysphagia after stroke: incidence, diagnosis, and pulmonary complications. Stroke. 2005 Dec;36(12):2756-63. doi: 10.1161/01.STR.0000190056.76543.eb. Epub 2005 Nov 3. PMID 16269630
- [Background] Chiara T, Martin AD, Davenport PW, Bolser DC. Expiratory muscle strength training in persons with multiple sclerosis having mild to moderate disability: effect on maximal expiratory pressure, pulmonary function, and maximal voluntary cough. Arch Phys Med Rehabil. 2006 Apr;87(4):468-73. doi: 10.1016/j.apmr.2005.12.035. PMID 16571384
- [Background] Kulnik ST, Birring SS, Moxham J, Rafferty GF, Kalra L. Does respiratory muscle training improve cough flow in acute stroke? Pilot randomized controlled trial. Stroke. 2015 Feb;46(2):447-53. doi: 10.1161/STROKEAHA.114.007110. Epub 2014 Dec 11. PMID 25503549